CLINICAL TRIAL: NCT02328443
Title: Evaluation and Validation of Metabolic Markers for the Assessment of CYP3A Activity and Prediction of Drug-drug Interaction in Korean Healthy Subjects
Brief Title: Evaluation and Validation of Metabolic Markers for the Assessment of CYP3A Activity and Prediction of DDI
Acronym: CYP3A_weak
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Youn Cho, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CYP3A_weak
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: CYP3A; Metabolomics
MeSH Terms: interventions — Midazolam; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- midazolam alone (Experimental): midazolam administration alone
  Interventions: Drug: Midazolam
- midazolam and itraconazole (Experimental): Itraconazole 200 mg PO twice; midazolam iv single administration
  Interventions: Drug: Midazolam; Drug: itraconazole
- midazolam and rifampicin (Experimental): rifampicin 150 mg PO for 9 days administration, midazolam iv single administration
  Interventions: Drug: Midazolam; Drug: rifampicin

INTERVENTIONS:
Drug: Midazolam
  Other Names: Bukwang Midazolam, Korea
Drug: itraconazole
  Arms: midazolam and itraconazole
Drug: rifampicin
  Arms: midazolam and rifampicin

SUMMARY:
Evaluation and validation of metabolic markers for the assessment of CYP3A activity and prediction of drug-drug interaction in Korean healthy subjects.

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trials Center, Seoul National University Hospital on the day before dosing, and they were overnight-fasted from 10 p.m. of Day -1. Urine collection is scheduled drug 12 hour before and 24 hour after midazolam administration. Subjects will be dosed study drug via intravenous around at 9 a.m. of Day 1. Subjects performed scheduled procedures.

In period 2, Subjects will be admitted on Day 3-5. Subjects performed scheduled period 2 (Itraconazole co-administration phase, 2 times administration of itraconazole 200 mg), and period 3 (rifampicin 150 mg co-administration phase) procedure. Study participation was terminated on post-study visit (Day 23~35).

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 40 years of age, inclusive
* Weight: within 17-28 of Body Mass Index (BMI)
* Subject who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of hypersensitive reaction to medication (midazolam, itraconazole, rifampicin)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History or evidence of drug abuse
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
* Participation in clinical trials of any drug within 60 days prior to the participation of the study
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quantitation of endogenous metabolites | -12h-24h
  endogenous metabolite profiles such as steroids to predict CYP3A activity
Maximum plasma concentration and area under the cure from zero to last point | Time Frame: 0h, 10m, 20m, 30m, 45m, 1h, 2h, 3h, 4h, 6h, 8h, 12h
  Cmax, AUClast of midazolam